CLINICAL TRIAL: NCT03964311
Title: Risk for Short-term Adverse Events in Older Emergency Department Users: '' Emergency Room Evaluation and Recommendation '' Cohort Study Database
Brief Title: Risk for Short-term Adverse Events in Older Emergency Department Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-1726
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Older People; Health Care; Evaluations; Health Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Room Evaluation Tool (ER2) (Other): Patients who are 75 years and over, and who are brought to Emergency in stretchers will be evaluated based on the Emergency Room Evaluation Tool (ER2).
  Interventions: Other: Emergency Room Evaluation Tool (ER2)

INTERVENTIONS:
Other: Emergency Room Evaluation Tool (ER2) — Emergency Room Evaluation Tool represents a screening method that will be used at the Emergency by nurses. This tool evaluates the health conditions of all the patients who are 75 years and over.

SUMMARY:
This study evaluates the association between risk levels (i.e.; low, moderate and high) of Emergency Room Tool (ER2) and length of stay in older Emergency Room Tool (ER) users admitted to the medical or surgery wards of the Jewish General Hospital.

DETAILED DESCRIPTION:
The Emergency Room Tool (ER2) assessment can be used by Emergency Department nurses taking care of older Emergency Department (ED) users on stretcher, and that ER2 moderate and high risk levels is associated with long length of stay in Emergency Department and hospital as well as hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Being 75 years and over
* An unplanned Emergency Department visit and to be on a stretcher.

Exclusion Criteria:

-Being 74 years and less

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Short-term adverse events | In around 30 days
  By using the Emergency Room Evaluation Tool( ER2), we will indirectly evaluate the length of hospital stay. The calculation will be done in days and hours.

SECONDARY OUTCOMES:
Usability of assessment tool | 24 hours in Emergency
  Patients at Emergency Room will be valuated by using the Emergency Room Evaluation Tool(ER2). Based on the ER2 results, it would be evaluated the usability of the Emergency Room screening tool.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Launay CP, Galery K, Vilcocq C, Afilalo M, Beauchet O. Risk for short-term undesirable outcomes in older emergency department users: Results of the ER2 observational cohort study. PLoS One. 2021 Aug 11;16(8):e0249882. doi: 10.1371/journal.pone.0249882. eCollection 2021. PMID 34379629